CLINICAL TRIAL: NCT00627393
Title: High Dose Granulocyte Transfusions for the Treatment of Infection in Neutropenia: The RING Study (Resolving Infection in Neutropenia With Granulocytes)
Brief Title: Safety and Effectiveness of Granulocyte Transfusions in Resolving Infection in People With Neutropenia (The RING Study)
Acronym: RING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 557; U01HL072268 (NIH); HL072268; HL072291; HL072196; HL072248; HL072191; HL072305; HL072028; HL072072; HL072355; HL072283; HL072346; HL072331; HL072290
Record Dates: First submitted 2008-02-28; First posted 2008-03-03 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Neutropenia; Infection
Keywords: Granulocyte Transfusions
MeSH Terms: conditions — Neutropenia; Infections | interventions — Filgrastim

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive granulocyte transfusions in addition to standard antimicrobial therapy
  Interventions: Drug: Standard antimicrobial therapy; Biological: Granulocyte transfusions
- 2 (Active Comparator): Participants will receive standard antimicrobial therapy alone
  Interventions: Drug: Standard antimicrobial therapy
- 3 (Other): Participants will donate granulocytes after receiving a combination of two drugs, G-CSF and dexamethasone
  Interventions: Drug: G-CSF/dexamethasone; Device: Apheresis machine

INTERVENTIONS:
Drug: Standard antimicrobial therapy — Antimicrobial therapy is broadly defined as therapy within the standard of care for a particular infection and should be consistent within a given institution. Participants will undergo the recommended therapy for specific infections for 42 days.
  Arms: 1; 2
Biological: Granulocyte transfusions — Participants will receive one granulocyte transfusion per day until one of the following occurs: recovery from neutropenia, life-threatening toxicity, resolution or improvement of infection, or Day 42 after treatment. Granulocyte content of each transfusion is targeted to be at least 4 x 10^10 per collection (or proportionately less for participants less than 30 kg in weight).
  Arms: 1
Drug: G-CSF/dexamethasone — Twelve hours before each donation, participants will be injected with G-CSF and will take one dose of dexamethasone by mouth.
  Other Names: Neupogen
  Arms: 3
Device: Apheresis machine — Participants will undergo a procedure using an apheresis machine for granulocyte collection. The procedure will last 3 to 4 hours and will involve the drawing of blood from each arm, the separation of granulocytes from the red cells and plasma in the machine, and the return of the red cells and plasma to the participants.
  Arms: 3

SUMMARY:
Neutropenia, a condition characterized by an abnormally low number of infection-fighting white blood cells called neutrophils, commonly develops in people who have undergone chemotherapy or hematopoietic stem cell (HSC) transplantation. The severely reduced immunity of those with neutropenia can put them at risk of entry of life-threatening infections, making the implementation of treatments that increase white blood cell numbers important. Several studies have shown that the transfusion of donor granulocytes, a type of white blood cell that includes neutrophils, is effective in promoting the recovery of adequate numbers of granulocytes. However, granulocyte transfusions can cause side effects, and it is not known whether the success of the therapy outweighs the health risks of the side effects. This study will evaluate the safety and effectiveness of granulocyte transfusions in treating people with a bacterial or fungal infection during neutropenia.

DETAILED DESCRIPTION:
Thousands of people each year are hospitalized for neutropenia, which continues to cause substantial morbidity and mortality for those affected. Neutropenia is primarily caused by chemotherapy and various other cancer treatments, such as radiation therapy, biotherapy, and HSC transplantation. Signs and symptoms of neutropenia may include high fever, chills, sore throat, and diarrhea. In neutropenia, the number of neutrophils, a type of granulocyte, is greatly reduced, weakening the body's immune system and increasing the risk of infection. Therefore, a method to provide adequate numbers of functional granulocytes to people with neutropenia could be of greatest benefit for recovery. Administration of a combination of two drugs, granulocyte colony-stimulating factor (G-CSF) and dexamethasone, has been show to stimulate the body to produce a large number of granulocytes. Granulocyte transfusions obtained from donors who have received these two drugs may help people with low white blood cell counts fight infections until their own white blood cell counts recover. However, it is not clear whether the benefits of granulocyte transfusions outweigh the risks of side effects. This study will compare the safety and effectiveness of granulocyte transfusions with standard antimicrobial therapy versus the safety and effectiveness of standard antimicrobial therapy alone in increasing granulocyte numbers and in improving survival rates in people with bacterial or fungal infection during neutropenia.

Participation in the research portion of this study will last about 3 months. All participants who were not previously receiving treatment with standard antimicrobial therapy will begin therapy immediately upon study entry. Participants will then be assigned randomly to receive either granulocyte transfusion plus continued antimicrobial therapy or continued antimicrobial therapy alone. All participants will be monitored for a maximum of 42 days, during which they will provide information on medical history and ongoing status of antimicrobial therapy. Daily blood samples to measure white blood cell count will be obtained from participants until samples show that participants are making their own granulocytes. Samples will then be collected weekly until Day 42. There may be additional blood draws depending on the type of infection present in participants.

Granulocyte transfusions will be given daily during the 42-day treatment period, depending on granulocyte donor availability. Blood counts will be checked immediately before and after each transfusion to measure granulocyte levels. Transfusions will be stopped if participants start making their own granulocytes, experience serious side effects, or show a reduction in infection. At Month 3 after study entry, follow-up information will be collected about all participants' health status through reviewing their medical records and contacting their physicians.

Participation for granulocyte donors will last 1 week from the time of donation. Community donors may provide more than one granulocyte donation, but no more than one donation every 3 days. Frequency of donation from a family member will be according to local blood bank criteria with approval from a blood bank physician. Both community donors and family donors are limited to eight donations each year. Twelve hours before each donation, participants will be injected with Neupogen, which contains G-CSF, and they will take one dose of dexamethasone by mouth. Participants will then undergo a blood draw, followed by a procedure using an apheresis machine for granulocyte collection. The procedure will last 3 to 4 hours and will involve the drawing of blood from each arm, the separation of granulocytes from the red blood cells and plasma in the machine, and the return of the red blood cells and plasma to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Severe neutropenia (Absolute Neutrophil Count < 500/mm^3) due to marrow failure caused by underlying disease or therapy
* Must have one of the following: fungemia; bacteremia; proven or presumptive invasive tissue bacterial infection; or proven, probable, or presumptive invasive fungal infection

Exclusion Criteria:

* Unlikely to survive 5 days
* Evidence that patient will not be neutropenic at least 5 days
* Previously enrolled in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-04; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F. Assmann, PhD, Principal Investigator — Carelon Research; Jan McFarland, MD, Principal Investigator — Froedtert Hospital; Eliot Williams, MD, Principal Investigator — University of Wisconsin, Madison; Ellis Neufeld, MD, Principal Investigator — Children's Hospital Boston/Brigham and Women's Hospital; James Bussel, MD, Principal Investigator — Weill Medical College, Cornell University; Cassandra Josephson, MD, Principal Investigator — Emory University; Paul Ness, MD, Principal Investigator — Johns Hopkins University; Sherrill Slichter, MD, Principal Investigator — University of Washington; Thomas Price, MD, Study Chair — Bloodworks; Ronald Strauss, MD, Principal Investigator — University of Iowa; Jeffrey McCullough, MD, Principal Investigator — University of Minnesota; James George, MD, Principal Investigator — University of Oklahoma; Bruce Sachais, MD, PHD, Principal Investigator — University of Pennsylvania; David Friedman, MD, Principal Investigator — Children's Hospital of Philadelphia; Darrell Triulzi, MD, Principal Investigator — University of Pittsburgh Presbyterian and Shadyside/Children's Hospital Pittsburgh
Locations (13):
- United States (13):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Medical College, Cornell University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Chlidren's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Presbyterian and Shadyside, Pittsburgh, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin at Madison, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Price TH, Boeckh M, Harrison RW, McCullough J, Ness PM, Strauss RG, Nichols WG, Hamza TH, Cushing MM, King KE, Young JA, Williams E, McFarland J, Holter Chakrabarty J, Sloan SR, Friedman D, Parekh S, Sachais BS, Kiss JE, Assmann SF. Efficacy of transfusion with granulocytes from G-CSF/dexamethasone-treated donors in neutropenic patients with infection. Blood. 2015 Oct 29;126(18):2153-61. doi: 10.1182/blood-2015-05-645986. Epub 2015 Sep 2. PMID 26333778

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: Received antimicrobial therapy alone.
- Granulocyte Arm: Received G-CSF/dexamethasone-mobilized granulocyte transfusions in addition to antimicrobial therapy.
Period: Intention-To-Treat Analysis
Arm/Group | Control Arm | Granulocyte Arm
Started | 58 | 56
Completed | 49 | 48
Not Completed | 9 | 8
Not completed — Adjudication indeterminate | 5 | 3
Not completed — Withdrawal by patient/family/physician | 4 | 5
Period: Per-Protocol Analysis
Arm/Group | Control Arm | Granulocyte Arm
Started | 49 | 48
Completed | 39 | 35
Not Completed | 10 | 13
Not completed — Received unstimulated/no granulocytes | 6 | 3
Not completed — Withdrawal by patient/family/physician | 4 | 10

BASELINE CHARACTERISTICS:
Population: All randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Granulocyte Arm | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 10
  Between 18 and 65 years | 39 | 32 | 71
  >=65 years | 13 | 20 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (19.8) | 54.8 (16.3) | 51.9 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 30 | 33 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 40 | 44 | 84
  Unknown or Not Reported | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 39 | 40 | 79
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 13 | 9 | 22
Weight [Mean (Standard Deviation); unit: kg] | 76.0 (23.8) | 78.7 (20.6) | 77.3 (22.2)
Cause of neutropenia [Number; unit: participants]
  Chemotherapy only | 43 | 44 | 87
  Infection | 7 | 3 | 10
  HST (or preparation for HST) | 8 | 9 | 17
ANC prior to randomization [Mean (Standard Deviation); unit: x10^9 cells/L] — ANC = Absolute neutrophil count.
  Subjects with ANC less than 500/mm^3 were considered to have severe neutropenia.
  x10^9 cells/L | 0.046 (0.091) | 0.058 (0.096) | 0.052 (0.094)
Zubrod score [Number; unit: participants] — The Zubrod scoring system ranks patients on their functionality on a scale from 0-5. Zubrod score category "0 to 2" represents asymptomatic, symptomatic but completely ambulatory, or symptomatic and 50% in bed during the day. Zubrod score category "3 to 5" represents symptomatic and more than 50% in bed (but not bedbound), being bedbound or completely disabled, or being moribund.
  participants
    0 to 2 | 19 | 18 | 37
    3 to 5 | 39 | 38 | 77
Infection type [Number; unit: participants]
  Bacteremia only | 16 | 17 | 33
  Tissue bacterial infection | 15 | 13 | 28
  Fungemia only | 8 | 5 | 13
  Tissue fungal infection | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Alive at 42 Days After Treatment and Have Had Microbial Response
Description: Microbial response was defined as follows:
  * A negative blood culture test at 42 days after randomization for subjects with fungemia (candidemia or fusariosis) or bacteremia.
  * Improvement of signs and symptoms of infectious disease (complete or partial response) at 42 days after randomization.
Time Frame: Measured at Day 42
Population: All adjudicated or deceased subjects in intention-to-treat analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm | Granulocyte Arm
Number analyzed (Participants) | 49 | 48
percentage of participants | 42.9 | 41.7
Statistical Analysis 1: Comparison: Control Arm vs Granulocyte Arm; Test type: Superiority or Other; p = 0.73, Regression, Logistic; Ordinary multiple logistic regression including treatment arm, infection strata, underlying disease, zubrod score, respiratory symptoms, and age; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.44 to 3.20] — Control group is the reference group. Model adjusted for infection strata, underlying disease, zubrod score, respiratory symptoms, and age

2. Secondary Outcome: Alloimmunization, Defined as the Appearance of Anti-human Leukocyte Antigen (HLA) or Antineutrophil Antibodies
Time Frame: Measured at Days 14 and 42
Reporting Status: Not Posted

3. Secondary Outcome: Serious Granulocyte Transfusion Reactions, Including Febrile, Allergic, and Pulmonary Reactions (Transfusion Arm Only)
Time Frame: Measured within 6 hours after end of transfusion
Population: Subjects who received granulocyte transfusions. Six subjects in the control group received granulocyte transfusions in violation of the protocol.
Measure: Number; unit: participants
Arm/Group | Control Arm | Granulocyte Arm
Number analyzed (Participants) | 6 | 51
participants
  No events reported | 5 | 19
  Grade 1 | 0 | 7
  Grade 2 | 1 | 14
  Grade 3 | 0 | 10
  Grade 4 | 0 | 1

4. Secondary Outcome: Graft Versus Host Disease Among Recipients of Allogeneic Stem Cell Transplantation
Description: Time to GVHD incidence between the two treatment groups was compared using Gray's model that takes into account death as a competing risk.
Time Frame: Measured at Day 42
Population: Subjects who had allogeneic stem cell transplantation
Measure: Number; unit: proportion of subjects, GVHD incidnence
Arm/Group | Control Arm | Granulocyte Arm
Number analyzed (Participants) | 8 | 7
proportion of subjects, GVHD incidnence | 0.67 | 0.40
Statistical Analysis 1: Comparison: Control Arm vs Granulocyte Arm; Test type: Superiority or Other; p = 0.43, Competing Risks — Competing risks analysis for time to GVHD for subjects with allogeneic HST. The sample size was very small (n=7 in the granulocyte group, and n=8 in the control group); Log Rank P-Value = 0.43

5. Secondary Outcome: Overall Incidence of Adverse Effects
Time Frame: Measured through Day 42
Population: All randomized subjects.
Measure: Number; unit: participants
Arm/Group | Control Arm | Granulocyte Arm
Number analyzed (Participants) | 58 | 56
participants
  0 Event | 33 | 30
  1 Event | 21 | 20
  2 Events | 2 | 5
  3 Events | 1 | 0
  6 Events | 0 | 1
  9 Events | 1 | 0

6. Secondary Outcome: Fever Resolution
Description: Fever resolution between the two treatment groups was compared using Gray's model that takes into account death as a competing risk.
Time Frame: Measured through Day 42
Population: Subjects who had fever at baseline.
Measure: Number; unit: proportion of subjects, resolved fever
Arm/Group | Control Arm | Granulocyte Arm
Number analyzed (Participants) | 53 | 47
proportion of subjects, resolved fever | 0.89 | 0.94

7. Secondary Outcome: Time to Negative Test for Fungal Antigenemia (e.g., Galactomannan Antigenemia Among Participants With Invasive Aspergillosis)
Time Frame: Measured at Days 7, 14, and 42
Reporting Status: Not Posted

8. Secondary Outcome: Time to Negative Blood Culture for Participants With Positive Blood Culture at Baseline
Time Frame: Measured through Day 42
Reporting Status: Not Posted

9. Secondary Outcome: Long-term Survival
Time Frame: Measured at Month 3
Population: All randomized subjects.
Measure: Number; unit: participants
Arm/Group | Control Arm | Granulocyte Arm
Number analyzed (Participants) | 58 | 56
participants | 30 | 20
Statistical Analysis 1: Comparison: Control Arm vs Granulocyte Arm; Test type: Superiority or Other; p = 0.35, Log Rank; Log-rank test to compare survival distributions between the control group and treatment group; Hazard Ratio (HR) = 1.293, 95% CI 2-sided [0.778 to 2.147], Standard Error of Mean 0.25885 — The control group is considered the reference group

10. Secondary Outcome: Serious Adverse Events in Granulocyte Donors
Time Frame: Measured at Week 1 after G-CSF administration
Population: 237 subjects consented to G-CSF and dexamethasone administration prior to granulocyte donation.
Measure: Number; unit: participants
Groups:
- Granulocyte Donors: Participants will donate granulocytes after receiving a combination of two drugs, G-CSF and dexamethasone
  G-CSF/dexamethasone: Twelve hours before each donation, participants will be injected with G-CSF and will take one dose of dexamethasone by mouth.
  Apheresis machine: Participants will undergo a procedure using an apheresis machine for granulocyte collection. The procedure will last 3 to 4 hours and will involve the drawing of blood from each arm, the separation of granulocytes from the red cells and plasma in the machine, and the return of the red cells and plasma to the participants.
Arm/Group | Granulocyte Donors
Number analyzed (Participants) | 237
participants
  Myalgia and backpain of unexpected duration | 1
  Abnormal nucleated red blood cell differential | 1

11. Secondary Outcome: Donor Availability (Proportion of Scheduled Granulocyte Transfusion Days on Which Granulocytes Were Available)
Time Frame: Measured through study completion
Population: The unit of analysis is patient-days where a granulocyte transfusion was scheduled.
Measure: Number; unit: percentage of available granulocyte days
Units Other Than Participants: Patient-days
Arm/Group | Granulocyte Arm
Number analyzed (Participants) | 56
Number analyzed (Patient-days) | 543
percentage of available granulocyte days | 62.62

12. Secondary Outcome: Evaluation of Granulocyte Yield
Time Frame: Measured immediately after each granulocyte donation
Measure: Median (Inter-Quartile Range); unit: Granulocyte Yield (billion cells/liter)
Units Other Than Participants: Granulocyte Donations
Arm/Group | Granulocyte Donors
Number analyzed (Participants) | 237
Number analyzed (Granulocyte Donations) | 340
Granulocyte Yield (billion cells/liter) | 174.75 [89.76 to 242.41]

13. Secondary Outcome: Discontinuation of Granulocyte Transfusions Due to Toxicity or Intolerance
Time Frame: Measured through Day 42
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious adverse events were reported up to 42 days after randomization.
Description: Serious adverse events and other adverse events (i.e. granulocyte transfusion related events) data were collected. The number of participants at risk for other adverse events corresponds to the number of participants who received granulocyte transfusions (6 control arm subjects and 51 granulocyte arm subjects).
Arm/Group | Control Arm | Granulocyte Arm
Serious Adverse Events (participants affected / at risk) | 25/58 | 26/56
Other Adverse Events (participants affected / at risk) | 1/6 | 32/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=58) | Granulocyte Arm (N=56)
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 2
Abdominal symptom (Gastrointestinal disorders) | 0 | 1 — Nausea, vomiting and abdominal pain.
Activated partial thromboplastin time shortened (Blood and lymphatic system disorders) | 1 | 0 — PTT (Grade 2)
Acute lung injury (Injury, poisoning and procedural complications) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Increased blast cell count (Blood and lymphatic system disorders) | 1 | 0
Increased blood creatinine (Blood and lymphatic system disorders) | 1 | 0
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Encephalopathy (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Fungaemia (Infections and infestations) | 2 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 1
Hallucination (General disorders) | 1 | 0
Hydraemia (Blood and lymphatic system disorders) | 0 | 1
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 1 | 0
Hypoalbuminaemia (Blood and lymphatic system disorders) | 1 | 0
Hypocalcaemia (Blood and lymphatic system disorders) | 1 | 0
Hypokalaemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Hypotension (General disorders) | 0 | 2
Infection in an immunocompromised host (Infections and infestations) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Multi-organ failure (General disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 0 | 1
Pelvic abscess (Reproductive system and breast disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased prothrombin level (Blood and lymphatic system disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sepsis neonatal (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Sepsis syndrome (Blood and lymphatic system disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=6) | Granulocyte Arm (N=51)
Allergic reaction/ hypersensitivity (Immune system disorders) | 0 (0) | 5 (5)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (3) | 17 (36)
Hypertension (General disorders) | 1 (1) | 9 (15)
Hypotension (General disorders) | 0 (0) | 10 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (16)
Headache (General disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Rigors and Chills (Musculoskeletal and connective tissue disorders) | 0 (0) | 15 (42)
Fever (General disorders) | 1 (2) | 28 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications and presentations resulting from studies from the TMH Network must be approved by the Publications and Presentations Committee before submission. The Sponsor (NERI) and funding agency (NHLBI) both are represented on the P&P Committee along with Network Investigators. Members of the P&P Committee can recommend changes to publications.